CLINICAL TRIAL: NCT05378711
Title: Evaluating the Results of Physician and Parent Decisions to Treat Selective Mutism With Fluoxetine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Jed Magen, Chair - Department of Psychiatry, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13-718F
Record Dates: First submitted 2014-05-19; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Selective Mutism; Social Anxiety
Keywords: Selective Mutism; Social Anxiety; Children; Adolescents
MeSH Terms: conditions — Mutism | interventions — Fluoxetine

STUDY DESIGN:
Masking Description: Participants serve as their own controls by being randomly assigned to switch from placebo to active medication at staggered start dates per single case design methodology.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoxetine (Experimental): Children will receive an introductory dose and therapeutic dose of fluoxetine at various time points in the study. Onset of fluoxetine is determined by assignment to a pre-determined randomized treatment schedule.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Children will receive a placebo or fluoxetine at different times dependent upon random assignment to a treatment schedule.
  Other Names: Prozac

SUMMARY:
The Department of Counseling, Educational Psychology, and Special Education and the Department of Psychiatry at Michigan State University have coordinated efforts to provide a diagnostic and treatment investigation for children, ages seven to eighteen, with Selective Mutism. The purpose of this study is to examine the utility of fluoxetine for the treatment of this debilitating disorder. Fluoxetine is expected to improve social anxiety and selective mutism symptomology.

DETAILED DESCRIPTION:
Children with selective mutism (SM) are at risk for current and continuing academic and socio-emotional difficulties. Unfortunately, this issue is complicated by the fact these children often respond poorly to psychosocial intervention. This leaves parents with the overwhelming decision to attempt a trial of medication regardless of the little available data on the evidence base of this approach. Despite the paucity of research, psychiatrists are prescribing fluoxetine for children with SM "off label", as the Food and Drug Administration (FDA) has yet to approve fluoxetine for this indication. This study blends the psychopharmacological expertise of psychiatrists with the mental health, systems, and psychological evaluation expertise of school psychologists to identify an appropriate psychopharmacological solution for children and adolescents with this debilitating disorder. To that end, this study will examine the utility of fluoxetine for the treatment of five children and adolescents, ages seven to eighteen, diagnosed with SM through the use of a non-concurrent multiple-baseline single-case design with a single-blind placebo-controlled procedure. Treatment effectiveness will be evaluated by visual analysis of the data, the Wampold and Worsham multiple-baseline design randomization test, and the Kendall's Tau + Mann-Whitney U effect size. Multiple methods of assessment including standardized measures, such as the Selective Mutism Questionnaire (SMQ), and behavior ratings, such as Direct Behavior Ratings (DBRs), will be used to gather baseline and treatment data. Multiple informants (i.e., parents, teachers, and psychiatrists) will provide information on treatment effect across settings (i.e., school and community). Information regarding adverse effects associated with fluoxetine treatment including a measure of behavioral disinhibition, parental acceptance of the fluoxetine intervention, and compliance with taking the medication will also be gathered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female from seven to seventeen years of age at their last birthday
* Meet DSM-IV-TR criteria for selective mutism
* No history of medication treatment for selective mutism
* Child has an immediate biological family member who is diagnosed with an anxiety disorder or has experienced symptoms of an anxiety disorder at some point in time
* Child has received 10 weeks of an evidence-based psychosocial treatment
* Child has never had a negative reaction to a psychopharmacological medication
* Child exhibits symptoms of social anxiety

Exclusion Criteria:

* Child is diagnosed with a speech condition, mental retardation, pervasive developmental disorder, or schizophrenia
* Child is an English language learner or from a different culture than the culture predominately represented within his or her school
* Child is taking or has taken any kind of a psychopharmacological medication (e.g., SSRI, MAO-I, stimulant, etc.)
* Child has a medical illness that may be complicated through the use of a psychopharmacological treatment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Selective Mutism Questionnaire (Change Over 15 Weeks) | 2 times per week for 15 weeks

SECONDARY OUTCOMES:
Multidimensional Anxiety Scale for Children - 2nd Edition (Change Over 15 Weeks) | 2 times per week for 15 weeks
Direct Behavior Ratings - Parent (Change Over 15 Weeks) | Parent (3 times per week for 15 weeks); Teacher (5 times per week for 15 weeks)
Clinical Global Impression (Change Over 15 Weeks) | Parent and Teacher (2 times per week for 15 weeks); Psychiatrist (biweekly for 15 weeks)
Side Effects Form for Children and Adolescents - Adapted (Change Over 15 Weeks) | biweekly for 15 weeks
Parent - Young Mania Rating Scale (Change Over 15 Weeks) | 2 times per week for 15 weeks
Treatment Evaluation Questionnaire - Parent | End of Study (after 15 weeks)

OTHER OUTCOMES:
Treatment Integrity Form | Daily for 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jed Magen, DO, Principal Investigator — Michigan State University; John Carlson, PhD, Principal Investigator — Michigan State University; Justin Barterian, MA, Principal Investigator — Michigan State University; Joel Sanchez, MD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University Psychiatry Clinic, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No